CLINICAL TRIAL: NCT01954901
Title: Hyperbaric Oxygen for Wagner II Diabetic Lower Extremity Ulcers: a Double-blind, Randomized,Controlled Clinical Trial.
Brief Title: Hyperbaric Oxygen for Wagner II Diabetic Lower Extremity Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to enroll subjects due to change in referral policy.
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDG20120029H
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Wagner Grade 2 Lower Extremity Ulcers
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard treatment plus Hyperbaric Oxygen (Experimental): The study treatment group will be compressed on air in the hyperbaric chamber to 2.0 atmospheres absolute (ATA), then placed on 100% oxygen by a head tent for 90 minutes.
  Interventions: Device: Hyperbaric oxygen therapy
- Standard treatment with Hyperbaric Room Air (Placebo Comparator): The study control group will be compressed to 2.0 ATA on air, then breath 21% oxygen and 79% nitrogen through the hood for 90 minutes.
  Interventions: Device: Hyperbaric room air

INTERVENTIONS:
Device: Hyperbaric oxygen therapy
  Arms: Standard treatment plus Hyperbaric Oxygen
Device: Hyperbaric room air
  Arms: Standard treatment with Hyperbaric Room Air

SUMMARY:
The purpose of this proposed DoD study is to determine if hyperbaric oxygen therapy (HBOT) plus standard wound care is more effective than standard wound care alone in the rate of healing and prevention of major amputation (metatarsal and proximal) in Wagner grade 2 diabetic lower extremity ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18.
2. Type 1 or 2 diabetes mellitus.
3. Wagner Grade 2 wound for at least 4 weeks. A diagnosis of a Wagner Grade 2 wound necessitates a persistent wound of 4 weeks (5).
4. DoD Beneficiary.

Exclusion Criteria:

1. Impending/urgent amputation due to ongoing or exacerbated infection.
2. Severe depression.
3. Claustrophobia.
4. Seizure disorder.
5. Uncontrolled asthma/severe COPD with pCO2 > 45 mmHg on arterial blood gas.
6. Grade 4 congestive heart failure.
7. Unstable angina.
8. Chronic/acute otitis media/sinusitis.
9. Major tympanic membrane trauma.
10. Prior chemotherapy with Bleomycin and evidence of deterioration in diffusing capacity after a single hyperbaric oxygen exposure.
11. Candidates for vascular surgery/angioplasty/stenting or patients with major large vessel disease. These patients could have peripheral vascular disease of such severity that hyperbaric treatment would not improve their condition.
12. Vascular surgery/angioplasty within the last 3 months. This exclusion controls for improvements to a patients vasculature and perfusion that occur within 1-2 months after vascular surgery/angioplasty. This will ensure that any perfusion changes to the patient's diabetic wound ulcer area recorded during the study are a result of hyperbaric therapy instead of recent vascular procedures.
13. Women who are breast feeding or of childbearing potential.
14. Dementia or mental disability rendering the potential subject incapable of following instructions or consenting to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes in wound size - wounds measured by length, width and depth | 14 months
Number of wounds healed | 14 months
Number of major and minor amputations | Three Years after initiation of study

SECONDARY OUTCOMES:
Peri-wound TCOM values | 14 months
Recurrence of ulceration | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: John B Slade, MD, Principal Investigator — David Grant Medical Center
Locations (1):
- David Grant USAF Medical Center, Travis Air Force Base, California, United States